CLINICAL TRIAL: NCT05940688
Title: Providing an Optimized and emPowered Pregnancy for You (PᵌOPPY) Feasibility Study
Acronym: PᵌOPPY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Heart Association (Other); ConnectionHealth (Unknown); Memora Health (Unknown)
Responsible Party: Principal Investigator, Rachel Sinkey, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 300009897; 22HERNPMI985239 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2023-06-25; First posted 2023-07-11 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Pregnancy; Infants; Disparities
Keywords: Pregnancy outcomes; Health inequities
MeSH Terms: interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: Study is a pilot randomized trial (n=40) randomizing eligible participants to usual care (n=10), or usual care plus a digital health intervention (n=10), or usual care plus a community health worker intervention (n=10), or usual care plus both a digital health intervention and a community health worker intervention.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Digital Health Intervention (Experimental): This group will receive routine prenatal care services. Additionally, those randomized to this arm will receive a DHI intervention. A modified DHI will be utilized that was developed by Memora Health in conjunction with EQUATE partners at UPenn and feedback from the POPPY Study Team and Community Advisory Board. All content is designed for 7th grade Flesch-Kincaid level or lower.
  Interventions: Behavioral: Digital Health intervention
- Community health worker (CHW) (Experimental): Individuals randomized to this group will receive routine prenatal care services. Additionally, they will receive a CHW intervention. The CHW intervention will be adapted from an ongoing CHW program in Jefferson County, AL called "From Day One (FDO)", a comprehensive patient-centered program designed to educate and provide non-clinical, psychosocial, emotional support to expectant mothers from the 1st trimester of pregnancy through their child's first year of life. The intervention has been modified by the POPPY Study Team and Community Advisory Board.
  Interventions: Behavioral: Community Health Worker
- DHI Plus CHW (Experimental): This group will receive routine prenatal care services. Additionally, this group will receive both DHI and CHW interventions.
  Interventions: Behavioral: Digital Health Intervention plus Community Health Worker
- Usual Care (No Intervention): This group will receive routine prenatal care services.

INTERVENTIONS:
Behavioral: Digital Health intervention — Health care information delivered via a link in a text message that is then opened in a secure browser.
  Other Names: DHI
  Arms: Digital Health Intervention
Behavioral: Community Health Worker — Health care information delivered via CHW.
  Other Names: CHW
  Arms: Community health worker (CHW)
Behavioral: Digital Health Intervention plus Community Health Worker — Health care information delivered via DHI plus CHW
  Arms: DHI Plus CHW

SUMMARY:
The P3OPPY Project is one of five projects within the American Heart Association P3 EQUATE Network. The overarching goal of the P3 EQUATE American Heart Association Health Equity Research Network (HERN) is to promote equity in Maternal and Infant Health outcomes by identifying innovative and cost-effective strategies to enhance access to quality health information, care, and experiences during pregnancy, postnatal and postpartum/preconception periods, particularly for Black and under-served populations. Collectively, the investigators will collaborate with pregnant and postpartum individuals and their families, hospitals, and communities to discover ways to reduce racism and social problems that contribute to poor health outcomes.

DETAILED DESCRIPTION:
Feasibility Study Aims

1. To assess the feasibility of the digital health (DHI) and community health worker (CHW) interventions by assessing participant acceptance and use of the intervention.
2. To assess study enrollment to determine appropriateness and usefulness of the inclusion and exclusion criteria to estimate enrollment duration in the planned trial.
3. To determine the number of prenatal visits and the incidence of some of the maternal and neonatal outcomes (ones with higher prevalence) or surrogate outcomes that will be targeted in the planned factorial design randomized controlled trial. (Data will be collected on all relevant maternal and neonatal outcomes. The randomized feasibility design will allow for effect size estimates of the intervention on the incidence of maternal and neonatal outcomes, which will aid in determining the appropriate target outcomes as well as power calculation of the more definitive trial.)

The PᵌOPPY study is designed to support the American Heart Association's mission to improve maternal/infant health outcomes and address inequities in maternal/infant health care. The promise of digital health and community health worker engagement makes PᵌOPPY interventions potentially transformative, sustainable, and scalable for Non-Hispanic Black mothers and their infants from under-served communities in Alabama and beyond. The objective of this pilot study is to determine if it is feasible to randomize and implement digital health and community health worker interventions.

Design Summary

The investigators will challenge existing care paradigms by testing the effectiveness of integrating innovative platforms into the existing healthcare system, including existing digital health and community health worker programs from within the EQUATE consortium, to eliminate critical barriers to equitable healthcare access. After seeking input from a Community Advisory Board, these interventions will be refined and deployed for pilot testing. Individuals in Non-Hispanic Black communities at the highest risk of adverse pregnancy outcomes which were historically underrepresented in clinical research due to structural racism will be included. The investigative team employs experts across the community, maternal, and infant health continuum.

For this pilot, 40 eligible participants will be randomized, 10 to usual care, 10 to DHI, 10 to CHW, and 10 to DHI + CHW

ELIGIBILITY:
Inclusion Criteria:

* Self Identifies as Non-Hispanic Black
* Between 16-49 years old
* Pregnant individuals between 8⁰ - 22⁶ weeks gestational age
* Live singleton or dichorionic twin gestation
* Dating sonogram at <23 weeks gestation
* Area Deprivation Index (ADI) National 4th or 5th Quintile
* Planning to deliver at UAB Hospital
* Speaks and writes in English
* No indication for delivery at the time of enrollment

Exclusion Criteria:

* Declines randomization
* Speaks or writes in languages other than English
* Currently incarcerated
* Fetal demise diagnosed prior to enrollment
* Known major structural chromosomal abnormalities prior to enrollment

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Sinkey, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Digital Health Intervention (DHI): This group will receive routine prenatal care services. Additionally, those randomized to this arm will receive a DHI intervention. A modified DHI will be utilized that was developed by Memora Health in conjunction with EQUATE partners at UPenn and feedback from the POPPY Study Team and Community Advisory Board. All content is designed for 7th grade Flesch-Kincaid level or lower.
Period: Overall Study
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Started | 9 | 10 | 11 | 10
Completed | 8 | 8 | 11 | 9
Not Completed | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care | Total
Number analyzed (Participants) | 9 | 10 | 11 | 10 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30.8 [23.5 to 34.0] | 29.5 [23.5 to 34.0] | 29.1 [23.5 to 34.0] | 24.9 [23.5 to 34.0] | 29.1 [23.5 to 34.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 11 | 10 | 40
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 9 | 10 | 11 | 10 | 40
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 10 | 11 | 10 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Participant Acceptance of Randomization Arm / Intervention
Description: Participant acceptance is defined as a yes response to this question:
  "I would recommend the care I received to someone in a similar situation."
Time Frame: 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants
  Yes | 8 | 8 | 10 | 7
  Missing or Unknown | 1 | 2 | 1 | 2
  No | 0 | 0 | 0 | 1

2. Primary Outcome: Participant Use of Digital Health and/or Community Health Worker Interventions
Description: Use of the intervention for the digital health arm(s) is defined as the % of opened text messages. Use of the intervention for the community health worker arm(s) is defined as the % of planned sessions in which the participant engages with the community health worker.
Time Frame: From randomization to 6 weeks postpartum
Population: We did not collect data for this outcome as planned because the University legal department would not allow texting in the manner initially planned.
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Outpatient Perinatal Care Visits
Description: Number of perinatal care visits
Time Frame: Randomization to study completion (up to 34 weeks)
Measure: Median (Inter-Quartile Range); unit: Visits
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Visits | 13 [11 to 14] | 9.5 [6.5 to 11] | 9 [4.5 to 10.5] | 12 [10.5 to 12]

4. Secondary Outcome: Preterm Birth
Description: Delivery of a neonate at less than 37 weeks
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Health Intervention | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants
  Yes | 2 | 1 | 4 | 3
  No | 7 | 7 | 7 | 7
  Missing | 0 | 2 | 0 | 0

5. Secondary Outcome: Neonatal Birthweight
Description: Weight of neonate at birth
Time Frame: At birth
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
grams | 3160.0 [2980 to 3480] | 3150.0 [2843.75 to 3577.5] | 2815.0 [2690 to 2990] | 2920.0 [2740 to 3060]

6. Secondary Outcome: Cesarean Delivery
Description: Occurrence of a cesarean birth
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Health Intervention | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants
  Cesarean | 7 | 5 | 3 | 3
  Vaginal | 2 | 3 | 8 | 7
  Missing | 0 | 2 | 0 | 0

7. Secondary Outcome: Maternal Blood Transfusion
Description: Transfusion of blood products
Time Frame: At birth
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Health Intervention | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants
  Yes | 1 | 0 | 1 | 2
  No | 8 | 8 | 10 | 8
  Missing | 0 | 2 | 0 | 0

8. Secondary Outcome: Breastfeeding Intent
Description: Participant's self-reported intent of whether or not to express breast milk upon admission to the delivery-associated hospitalization
Time Frame: Upon admission to the delivery-associated hospitalization
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Health Intervention | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants
  Breastfeed only | 2 | 1 | 1 | 2
  Formula feed only | 3 | 3 | 3 | 1
  Both breast and formula feed | 3 | 1 | 1 | 6
  Do not know yet | 1 | 3 | 2 | 1
  Missing | 0 | 2 | 4 | 0

9. Secondary Outcome: Vaccination Rate
Description: The number of mothers who received Tdap and infants who received the Hep B vaccine.
Time Frame: Pregnancy through 6 weeks postpartum / 6 weeks of life
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants
  Maternal TDAP: Accepted | 7 | 4 | 5 | 5
  Maternal TDAP: Did not receive | 2 | 6 | 6 | 5
  Maternal TDAP: Newborn Death | 0 | 0 | 0 | 0
  Newborn Hep. B: Accepted | 6 | 6 | 6 | 7
  Newborn Hep. B: Did not receive | 3 | 3 | 5 | 3
  Newborn Hep. B: Newborn Death | 0 | 1 | 0 | 0

10. Secondary Outcome: Maternal Postpartum Readmission
Description: Admission of the mother to the hospital after discharge from the delivery-associated hospitalization
Time Frame: From discharge from the delivery-associated hospitalization to 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants
  Readmission | 0 | 0 | 1 | 2
  No Readmission | 9 | 10 | 10 | 8

11. Secondary Outcome: Neonatal Hospital Readmission
Description: Answer to the question " How is your baby doing?"
Time Frame: Birth to 6 weeks of life
Measure: Count of Participants; unit: Participants
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
Number analyzed (Participants) | 9 | 10 | 11 | 10
Participants
  Healthy | 8 | 8 | 7 | 7
  Some Illness (Hospitalization, Clinic, or ER) | 0 | 0 | 0 | 1
  Baby Died | 0 | 0 | 4 | 1
  Missing | 1 | 2 | 0 | 1

ADVERSE EVENTS:
Time Frame: Randomization to 6-weeks postpartum, up to 40 weeks
Arm/Group | Digital Health Intervention (DHI) | Community Health Worker (CHW) | DHI Plus CHW | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10 | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT05940688/Prot_SAP_000.pdf